CLINICAL TRIAL: NCT04757077
Title: The Association Between Pelvic Floor Muscle Function, Diastasis Recti and Postpartum Pelvic Girdle Pain - a Matched Case Control Study.
Status: Completed | Type: Observational
Sponsor: Żelazna Medical Centre, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: PN/54/2021
Record Dates: First submitted 2021-02-15; First posted 2021-02-16 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-04

CONDITIONS: Pelvic Girdle Pain; Diastasis Recti and Weakness of the Linea Alba; Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Girdle Pain; Diastasis Recti And Weakness Of The Linea Alba; Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GROUP 1: Patients 6-24 weeks after delivery with postpartum PGP (Patients with symptoms and signs of PGP, PGP confirmed with dedicated functional tests).
- GROUP 2: Patients 6-24 weeks after delivery, with no symptoms and signs of PGP.

SUMMARY:
Background: Pregnancy-related pelvic girdle pain (PGP) can appear during pregnancy, directly after labour or can be delayed to 3 weeks postpartum. Pain is experienced between the posterior iliac crest and the gluteal fold, particularly in the vicinity of the sacroiliac joint (SIJ). The pain may radiate in the posterior thigh and can also occur in conjunction with/or separately in the symphysis. The endurance capacity for standing, walking, and sitting is diminished. The diagnosis of PGP can be reached after exclusion of lumbar causes. The pain or functional disturbances in relation to PGP must be reproducible by specific clinical tests. Lack of accurate and early diagnosis of the PGP postpartum may contribute to development of chronic condition, lowering quality of life years after delivery. There is uncertainty regarding the association between the function of the pelvic floor muscles (PFM), diastasis recti and postpartum pelvic girdle pain (PGP). Although widely researched abroad, there is a paucity in research about biopsychosocial profile of women with postpartum PGP in Poland.

Objectives: The aim of this one-to-one matched case-control study it to examine whether there is any difference in PFM function and diastasis recti between women with and without clinically diagnosed PGP. Additionally, differences in biopsychosocial profile (depression, anxiety, stress, catastrophizing and kinesiophobia) will be assessed.

Materials and methods: Because of low incidence of researched condition, a case control study will be the study design of choice. Women 6-24 weeks after delivery with postpartum PGP will be matched with those with no PGP. Subjects' assessment will consist of palpation examination of diastasis recti (inter-recti distance) and pelvic floor muscles. Perineometry of the pelvic floor will also be conducted. Additionally, several questionnaires for the assessment of mental processing will be used: Depression Anxiety Stress Scale 21, Pain Catastrophizing Scale and Tampa Scale of Kinesiophobia. Participants will be matched according to age, parity and time postpartum.

Expected results: To our knowledge, postpartum pelvic girdle pain has not been extensively studied in Poland so far. The study will bring information about the possible associations with postpartum PGP. We hypothesize that the study will confirm our clinical observations about pelvic floor dysfunction and maladaptive mental processing in women with postpartum PGP.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal labour (including vacuum extractor or forceps) or caesarean section
* For group with PGP: pain due to PGP
* For control group with no pain - no pain due to PGP
* Agreement to participate

Exclusion Criteria:

* Diseases that can mimic PGP f.ex. Scheuermann disease, rheumatoid arthritis, Ehler's-Danlos Syndrome, hip dysplasia.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women, 6-24 weeks after delivery
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Perineometry of the pelvic floor - vaginal resting pressure. | one time assessment, 6-24 weeks after delivery
  Measurement of the vaginal resting pressure.
Perineometry of the pelvic floor - vaginal squeeze pressure. | one time assessment, 6-24 weeks after delivery
  Measurement of the vaginal squeeze pressure.
Palpable measurement of inter-recti distance (IRD) | one time assessment, 6-24 weeks after delivery
  Palpable measurement of inter-recti distance (IRD)

SECONDARY OUTCOMES:
Perineometry of the pelvic floor - endurance | one time assessment, 6-24 weeks after delivery
  Pelvic floor endurance measurement (area under the curve).
Diastasis Recti: palpation examination of the stability of the linea alba | one time assessment, 6-24 weeks after delivery
  Assesment of the stability of the linea alba during abdominal crunch - bulging means that it is unstable
Palpation examination of pelvic floor muscles with the use of PERFECT Scheme | one time assessment, 6-24 weeks after delivery
  Assesment of pelvic floor muscles with the use of PERFECT Scheme
Pain Catastrophizing Scale | one time assessment, 6-24 weeks after delivery
  Assesment of Catastrophizing. It consists of 13 items rated on 5- point scale (0-not at all, 4-all the time). The score range is 0-52. Higher scores indicates higher amounts of pain catastrophizing.
Depression Anxiety Stress Scale 21 | one time assessment, 6-24 weeks after delivery
  Assesment of Catastrophizing. It is a self-report scale which consists of 21 items and 4-point severity scales (0- did not apply to me at all, 3-applied to me very much, or most of the time). Total scale thus range between 0 and 120, and those for each of the subscales may range between 0 and 42. Moderate outcomes indicates elevated depression, anxiety, or stress.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Sophia's Specialist Hospital, Warsaw, Poland